CLINICAL TRIAL: NCT05924347
Title: Longitudinal MRI Study to Catch EARLY Scoliotic Changes of the Bone and Intervertebral Disc in Younger Sisters and Daughters of Adolescent Idiopathic Scoliosis Patients and the 22q11.2DS Population.
Brief Title: Early Scoliotic Changes in Children at Increased Risk for Scoliosis Development
Acronym: EARLYBIRD
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Eindhoven University of Technology (Other)
Responsible Party: Principal Investigator, dr. Tom P.C. Schlösser, Principal Investigator, UMC Utrecht
Other Study IDs: NL82419.041.22
Record Dates: First submitted 2023-01-26; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Adolescent Idiopathic Scoliosis; 22q11.2 Deletion Syndrome
MeSH Terms: conditions — DiGeorge Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: 60 adolescent girls (8-10 years old) at increased risk for idiopathic scoliosis development (an older sibling or parent diagnosed with idiopathic scoliosis)
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Scolioscan; Diagnostic Test: Skeletal maturity assessment
- Cohort 2: 60 adolescent girls or boys with the 22q11.2DS with increased risk for idiopathic-like scoliosis development.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Scolioscan; Diagnostic Test: Skeletal maturity assessment

INTERVENTIONS:
Diagnostic Test: MRI — Longitudinal MRI examination of the thoracic and lumbar spine (T2, T2w, sCT)
Diagnostic Test: Scolioscan — 3D ultrasound of the spine
Diagnostic Test: Skeletal maturity assessment — At one timepoint, a Hand radiograph is taken for digital skeletal maturity assessment

SUMMARY:
Rationale: Despite several decades of research, the exact etiology of adolescent idiopathic scoliosis (AIS) remains unclear. In AIS, spine curvature begins with and progresses during the adolescent growth spurt. Previous studies are only performed on populations with already established scoliosis and normal spinal growth (of bone and IVD tissue) during adolescence has also not been defined. Growth pattern differences may exist between scoliotic and nonscoliotic subjects. Previous studies support the hypothesis that AIS is a spinal deformity that starts with decompensation in the IVD and is linked to sagittal spinal alignment. However, to understand its cause and pathogenic mechanism, the changes to the adolescent spine must be assessed longitudinally during the growth period coinciding with the period prior to and during the onset of AIS. Ideally this should include a cohort who do and do not develop AIS and their assessment must be minimally harmful, without radiation exposure. Certain populations are at increased risk for scoliosis development (i.e. girls with family members with scoliosis and 22q11.2DS patients). New imaging modalities (boneMRI, 3D spinal ultrasound) allow for non-radiographic monitoring of spinal growth.

DETAILED DESCRIPTION:
Objective: The primary objectives is: To longitudinally evaluate the substantial differences in anatomical changes in the spine during adolescent growth in girls, at increased risk for scoliosis development, and in adolescent 22q11.2DS patients, that do and do not develop AIS.

The secondary objectives are:

* To develop spine specific (IVD/endplates) maturity assessment grading.
* To implement radiation-free imaging methods for spinal monitoring in adolescent patients at risk for scoliosis development.
* To create a longitudinal dataset for patient specific spinal biomechanical assessment.

Study design: Prospective observational cohort study

Study population: 60 adolescent girls (8-10 years old) at increased risk for idiopathic scoliosis development (an older sibling or parent diagnosed with idiopathic scoliosis) (Cohort-1) and 60 adolescent girls and boys with 22q11.2DS with increased risk for idiopathic-like scoliosis development (Cohort-2).

Intervention: none

Main study parameters/endpoints: Spinal MR imaging of the thoracic and lumbar spine will be performed at 5 time points between 8 or 9 and 15 or 16 for girls and boys respectively to evaluate possible changes in the 3D anatomy of the spine. The main study parameter will be the longitudinal changes in segmental axial rotation on boneMRI of the thoracolumbar spine in subjects that do and do not develop AIS.

Secondary endpoints: Changes in bone and intervertebral disc morphology, lateral shift of the nucleus pulposus. These will be correlated to assessments of growth, skeletal maturity and spinal alignment.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* Female,
* 8, 9 or 10 years old
* An older sibling, twin or parent diagnosed with AIS

Cohort 2:

* Diagnosed with 22q11.2DS
* Girls: 8, 9 or 10 years old.
* Boys: 9, 10 or 11 years old.

All

* No clinical signs of scoliosis at inclusion (physical examination by forward bending test and Bunnell Scoliometer assessment with a cut-off value of 7°.
* Written informed consent of parents/legal representatives.

Exclusion Criteria:

* Contraindications for MR imaging
* Early-onset scoliosis or other spinal deformities
* Other syndromes or neuromuscular disease associated with scoliosis
* Clinical signs of >1cm leg length discrepancy
* Other diseases or injuries, that are related to abnormal spinal growth, posture, activity levels, or scoliosis development.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cohort 1: 60 adolescent girls (8-10 years old) at increased risk for idiopathic scoliosis development (an older sibling or parent diagnosed with idiopathic scoliosis) Cohort 2: 60 adolescent girls or boys with the 22q11.2DS with increased risk for idiopathic-like scoliosis development.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2032-05 (Estimated); Study Completion 2032-05-01 (Estimated)

PRIMARY OUTCOMES:
Spinal MR Imaging of the thoracic and lumbar spine | Girls: Baseline
  MRI images
Spinal MR Imaging of the thoracic and lumbar spine | Girls: 11year
  MRI images
Spinal MR Imaging of the thoracic and lumbar spine | Girls: 12year
  MRI images
Spinal MR Imaging of the thoracic and lumbar spine | Girls: 13year
  MRI images
Spinal MR Imaging of the thoracic and lumbar spine | Girls: 15year
  MRI images
Spinal MR Imaging of the thoracic and lumbar spine | Boys: Baseline
  MRI images
Spinal MR Imaging of the thoracic and lumbar spine | Boys: 12year
  MRI images
Spinal MR Imaging of the thoracic and lumbar spine | Boys: 13year
  MRI images
Spinal MR Imaging of the thoracic and lumbar spine | Boys: 14year
  MRI images
Spinal MR Imaging of the thoracic and lumbar spine | Boys: 16year
  MRI images

SECONDARY OUTCOMES:
A-P ratio vertebrae and disc | Girls: Baseline
  Ratio anterior and posterior height
A-P ratio vertebrae and disc | Girls: 11year
  Ratio anterior and posterior height
A-P ratio vertebrae and disc | Girls: 12year
  Ratio anterior and posterior height
A-P ratio vertebrae and disc | Girls: 13year
  Ratio anterior and posterior height
A-P ratio vertebrae and disc | Girls: 15year
  Ratio anterior and posterior height
A-P ratio vertebrae and disc | Boys: Baseline
  Ratio anterior and posterior height
A-P ratio vertebrae and disc | Boys: 12year
  Ratio anterior and posterior height
A-P ratio vertebrae and disc | Boys: 13year
  Ratio anterior and posterior height
A-P ratio vertebrae and disc | Boys: 14year
  Ratio anterior and posterior height
A-P ratio vertebrae | Boys: 16year
  Ratio anterior and posterior height
Left-right ratio | Girls: Baseline
  Ratio left and right height
Left-right ratio | Girls: 11year
  Ratio left and right height
Left-right ratio | Girls: 12year
  Ratio left and right height
Left-right ratio | Girls: 13year
  Ratio left and right height
Left-right ratio | Girls: 15year
  Ratio left and right height
Left-right ratio | Boys: Baseline
  Ratio left and right height
Left-right ratio | Boys: 12year
  Ratio left and right height
Left-right ratio | Boys: 13year
  Ratio left and right height
Left-right ratio | Boys: 14year
  Ratio left and right height
Left-right ratio | Boys: 16year
  Ratio left and right height
Torsion | Girls: Baseline
  Difference in axial rotation between 2 subsequent endplates
Torsion | Girls: 11year
  Difference in axial rotation between 2 subsequent endplates
Torsion | Girls: 12year
  Difference in axial rotation between 2 subsequent endplates
Torsion | Girls: 13year
  Difference in axial rotation between 2 subsequent endplates
Torsion | Girls: 15year
  Difference in axial rotation between 2 subsequent endplates
Torsion | Boys: Baseline
  Difference in axial rotation between 2 subsequent endplates
Torsion | Boys: 12year
  Difference in axial rotation between 2 subsequent endplates
Torsion | Boys: 13year
  Difference in axial rotation between 2 subsequent endplates
Torsion | Boys: 14year
  Difference in axial rotation between 2 subsequent endplates
Torsion | Boys: 16year
  Difference in axial rotation between 2 subsequent endplates
Volumes disc | Girls: Baseline
  Volumes disc
Volumes disc | Girls: 11year
  Volumes disc
Volumes disc | Girls: 12year
  Volumes disc
Volumes disc | Girls: 13year
  Volumes disc
Volumes disc | Girls: 15year
  Volumes disc
Volumes disc | Boys: Baseline
  Volumes disc
Volumes disc | Boys: 12year
  Volumes disc
Volumes disc | Boys: 13year
  Volumes disc
Volumes disc | Boys: 14year
  Volumes disc
Volumes disc | Boys: 16year
  Volumes disc
Volumes vertebrae | Girls: Baseline
  Volumes vertebrae
Volumes vertebrae | Girls: 11year
  Volumes vertebrae
Volumes vertebrae | Girls: 12year
  Volumes vertebrae
Volumes vertebrae | Girls: 13year
  Volumes vertebrae
Volumes vertebrae | Girls: 15year
  Volumes vertebrae
Volumes vertebrae | Boys: Baseline
  Volumes vertebrae
Volumes vertebrae | Boys: 12year
  Volumes vertebrae
Volumes vertebrae | Boys: 13year
  Volumes vertebrae
Volumes vertebrae | Boys: 14year
  Volumes vertebrae
Volumes vertebrae | Boys: 16year
  Volumes vertebrae
Shift nucleus pulposis | Girls: Baseline
  Position of nucleus pulposus in discus
Shift nucleus pulposis | Girls: 11year
  Position of nucleus pulposus in discus
Shift nucleus pulposis | Girls: 12year
  Position of nucleus pulposus in discus
Shift nucleus pulposis | Girls: 13year
  Position of nucleus pulposus in discus
Shift nucleus pulposis | Girls: 15year
  Position of nucleus pulposus in discus
Shift nucleus pulposis | Boys: Baseline
  Position of nucleus pulposus in discus
Shift nucleus pulposis | Boys: 12year
  Position of nucleus pulposus in discus
Shift nucleus pulposis | Boys: 13year
  Position of nucleus pulposus in discus
Shift nucleus pulposis | Boys: 14y
  Position of nucleus pulposus in discus
Shift nucleus pulposis | Boys: 16year
  Position of nucleus pulposus in discus
Changes in spinal alignment during growth | Girls: Baseline-15years, Boys: Baseline-15years
  Scan for changes over growth
Spine specific maturity assessment grading | Girls: Baseline-15years, Boys: Baseline-15years
  See if it is possible to create a spine specific maturity assessment

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lafranca PPG, Stempels HW, de Reuver S, Houben ML, Kok J, Kruyt MC, Castelein RM, Seevinck PR, van der Velden T, Shcherbakova YM, Ito K, Schlosser TPC. EARLYBIRD: catching the earliest changes of the bone and intervertebral discs in children at increased risk for scoliosis development with MRI - study protocol of a prospective observational cohort study. BMJ Open. 2025 Jun 26;15(6):e098929. doi: 10.1136/bmjopen-2025-098929. PMID 40578865